CLINICAL TRIAL: NCT07308301
Title: EXAMİNATİON OF THE RELATİONSHİP BETWEEN QUALİTY OF LİFE AND CAREGİVİNG BURDEN AMONG CAREGİVERS OF PEDİATRİC OCOLOGY PATİENTS
Brief Title: Examination of the Relationship Between Quality of Life and Caregiving Burden Among Caregivers of Pediatric Oncology Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Fatma Beyza Akdeniz (Other)
Responsible Party: Sponsor-Investigator, Fatma Beyza Akdeniz, Pediatric Nurse, Fenerbahce University
Organization: Fenerbahce University (Other)
Other Study IDs: 2024-KAEK-11
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Childhood Cancer; Childhood Cancers; Caregiver Subjective Burden; Primary Caregivers of Children Newly Diagnosed With Cancer; Caregiver; Caregiver Anxiety; Caregiver Health Related QOL
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary caregivers eighteen and older of hospitalized pediatric cancer patients will be included.: The study includes individuals who provide care for pediatric oncology patients. The research will involve primary caregivers aged 18 years or older who provide care for a child diagnosed with cancer and who are currently hospitalized in the Pediatric Hematology and Oncology Unit of Başakşehir Çam and Sakura City Hospital. The study will examine caregivers' sociodemographic characteristics, quality of life, and caregiving burden levels.
  Interventions: Behavioral: Assessment of caregiver quality of life and burden

INTERVENTIONS:
Behavioral: Assessment of caregiver quality of life and burden — This intervention consists of assessing the quality of life and caregiving burden of primary caregivers of children diagnosed with cancer using standardized questionnaires and scales. It does not involve any medical procedures, treatments, or experimental applications. The intervention includes only the administration of data collection tools to caregivers and is therefore distinct from treatment-based interventions used in other clinical studies.

SUMMARY:
Primary Aim

The primary aim of this study is to determine the quality of life and caregiving burden levels of caregivers of pediatric oncology patients and to examine the relationship between these two variables.

Secondary Aims

To evaluate the differences between caregivers' sociodemographic characteristics (age, gender, education level, marital status, income level, etc.) and their quality of life.

To examine the differences between caregivers' sociodemographic characteristics and their caregiving burden levels.

To determine whether caregivers' quality of life and caregiving burden differ according to the diagnosis and treatment characteristics of pediatric oncology patients (duration of diagnosis, type of treatment, frequency of hospitalization, etc.).

Significance of the Study

Childhood cancer is a process that deeply affects not only the patient but also the family, particularly the caregivers. Family members who provide care for children often face intense physical, psychological, social, and economic burdens. These challenges reduce caregivers' quality of life and increase their caregiving burden.

Identifying the relationship between the quality of life and caregiving burden among caregivers of pediatric oncology patients is highly important in planning support services for families during the care process and in strengthening family-centered care practices by healthcare professionals.

The findings of this study will contribute to the development of family-centered approaches in nursing care, the design of psychosocial support programs, and a better understanding of caregivers' needs.

ELIGIBILITY:
Inclusion Criteria:

* Being a family member who provides care for a child aged 0-18 years diagnosed with cancer
* The child being in the active treatment phase (chemotherapy, radiotherapy, post-surgical follow-up, etc.)
* Being able to read and write in Turkish and having sufficient literacy to complete the research questionnaire
* Willingness to participate in the study

Exclusion Criteria:

* Not being the primary caregiver of the child (serving only as a short-term companion)
* Being unable to complete the questionnaire due to a psychiatric diagnosis or communication difficulties
* The child having a disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study includes individuals who provide care for pediatric oncology patients. Primary caregivers aged 18 years and older who provide care for children diagnosed with cancer and who are hospitalized in the Pediatric Hematology-Oncology Unit of Başakşehir Çam and Sakura City Hospital will be included in the study. The study will examine caregivers' sociodemographic characteristics, quality of life, and levels of caregiving burden.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Caregiver Quality of Life Index-Cancer (CQOLC) | From the enrollment phase until the end of the 12-week data collection period.
  The scale consists of 25 items and four subscales: burden (10 items: 9, 11, 14, 15, 18, 19, 20, 21, 25, 31), disruptiveness (6 items: 1, 2, 3, 5, 13, 29), positive adaptation (6 items: 17, 24, 26, 30, 32, 33), and financial distress (3 items: 6, 7, 8). The scale is rated on a Likert-type scale ranging from 0 (almost never), 1 (not much), 2 (somewhat), 3 (quite a bit), to 4 (very much).
  Subscale scores of the CQOLC are calculated by summing the items within each subscale. The total CQOLC score is obtained by summing all 25 items. The total CQOLC score ranges from 0 to 100, with higher scores indicating lower quality of life. The overall internal consistency coefficient of the scale is .88, while the Cronbach's alpha values for the subscales of burden, disruptiveness, positive adaptation, and financial distress are reported as .83, .79, .73, and .77, respectively.

SECONDARY OUTCOMES:
Caregiver Burden Scale | From the enrollment phase until the end of the 12-week data collection period.
  The scale consists of 36 items rated on a 5-point Likert scale and includes four subscales. The emotional burden subscale comprises 12 items, the sociocultural and economic burden subscale comprises 11 items, the mental burden subscale comprises 7 items, and the physical burden subscale comprises 6 items. Participants completing the scale indicate their level of agreement with statements related to the caregiving burden experienced during the process of caring for their child using the following response options: "1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Always." The minimum possible total score is 36 (36 items × 1 point), and the maximum possible total score is 180 (36 items × 5 points). The caregiver burden level is determined by summing the responses to all items. Accordingly, mean score ranges are interpreted as follows: mean scores of 1.00-2.00 indicate "no or low burden," 2.00-3.00 indicate "mild to moderate burden," 3.00-4.00-5.00 indicate "

IPD SHARING:
Plan to Share IPD: Undecided